CLINICAL TRIAL: NCT06804278
Title: Role of Spectral CT in the Diagnosis of Myocarditis/MINOCA in Patients Undergoing cardioCT Investigations for Acute Chest Pain
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MioSpectralCT
Record Dates: First submitted 2025-01-09; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Imaging Techniques; Cardiac Imaging; Myocardial Disease; Myocarditis Acute; Minoca
MeSH Terms: conditions — Cardiomyopathies; MINOCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a spontaneous, observational cross-sectional and single-center imaging (CT and MRI) study, coupled with clinical-laboratory data. Patients with acute chest pain with low/intermediate probability of coronary artery disease, ECG and/or troponin not diagnostic or altered according to the current "standards of care" used in the ED/Department (ESC Guidelines 2020), will be enrolled consecutively and will undergo CT examinations by means of "Spectral" CT technology. CT investigation will allow to identify any non-myocarditis causes of acute chest pain and by means of spectral analysis of CT images it will try to identify signs suggestive of damage myocardial (such as ECV, LIE, hyperemia and edema).

DETAILED DESCRIPTION:
Innovation in the field of CT (Computed Tomography) with the introduction of new technologies, including the detector-based SpectralCT or Spectral CT (SDCT), has led in recent years to a true "paradigm-shift" from an evaluation of CT images on a purely "observational" to the "radiomics" level, allowing the introduction of additional valuable quantitative information, obtained only through post-processing with software CT images. In particular, Spectral CT is a scanner dedicated to tissue characterization thanks to its ability to "break down" and separate the different materials that make up fabrics, creating sets of monoenergetic (different KeV) or selective (water, iodine, etc.) images.

With this method, it is therefore possible to obtain information previously obtainable with conventional CT equipment, such as iodine maps, medium subtraction tissue characterization data through the calculation of extracellular volume (ECV), the visualization of hyperemia, edema and much more. It is precisely the ability to characterize myocardial tissue, in particular to highlight edema or a fibrotic replacement by ECV calculation and late iodine enhancement (LIE), is one of the most interesting aspects of this new method in the field of imaging cardiovascular, for example in the urgent/emergency setting, where radiology plays a key role in the evaluation of the main causes of acute chest pain, such as heart attack, pulmonary embolism, acute aortic syndromes and myocarditis.

In particular, CT is the first-line method in patients with acute chest pain with low/intermediate probability of coronary artery disease, ECG and/or non-diagnostic troponin(s) or and has already demonstrated its ability to simultaneously exclude disease coronary artery, pulmonary embolism, and aortic dissection through a single examination commonly called "Triple rule out".

To date, however, the non-invasive diagnosis of myocarditis/MINOCA (Myocardial Infarction at coronary arteries) is not obtainable from the evaluation of conventional CT images and is prerogative of cardiac magnetic resonance imaging (MRI) [3]. The added value of the "Spectral CT", thanks to the characteristics described above, could be that of highlighting and/or excluding, in addition to the three aforementioned causes of acute chest pain (i.e. heart attack, pulmonary embolism and acute aortic syndrome), also acute myocarditis or MINOCA The new technology on which SpectralCT is based could in fact make it possible to highlight signs suggestive of myocardial damage, such as ECV, LIE, hyperemia and edema, by post-processing of the same CT images acquired in usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years;
* patients with acute chest pain and indication for triple-rule-out CT or coronary CT examination, i.e. low/intermediate probability of acute coronary artery disease, ECG and/or troponin not diagnostic or altered;
* Obtaining informed consent

Exclusion Criteria:

* Absolute contraindications to CT examination and/or iodinated mdc administration (i.e. pregnancy, severe renal impairment in non-dialysis patients with GFR < 15-30 ml/min/1.73m2 );
* CT examinations that do not allow diagnostic information to be provided because they are assessed as quality too scarce and not interpretable (affected by artifacts such as motion artifacts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients from ED or the other wards of the IRCCS University Hospital of Bologna (department of Cardiology Intensive Care, Cardiology Unit), with acute chest pain and low/intermediate probability of coronary artery disease, ECG and/or troponin not diagnostic or altered, which will be subjected to cardiac CT examinations using "Spectral" technology and possibly MRI examinations by the cardioradiology team of the Radiology Unit, IRCCS University Hospital of Bologna.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
number of myocarditis or MINOCA diagnosed with Spectral CT | 1 week after examination
  Diagnosis of the presence of myocarditis/MINOCA will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Russo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No